CLINICAL TRIAL: NCT05050981
Title: Comparison of Effects of Menopause Hormonal Therapy and Selective Serotonin Reuptake in Postmenopausal Women
Brief Title: Effects of Menopause Hormonal Therapy and Selective Serotonin Reuptake Inhibitor on Cognition, Sexual Function and Quality of Life
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Luciano de Melo Pompei', Auxiliary Professor at Gynecology Department, Faculdade de Medicina do ABC
Other Study IDs: 40147320.5.0000.0082
Record Dates: First submitted 2021-09-02; First posted 2021-09-21 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Menopause
Keywords: menopause; hormone replacement therapy; selective serotonin reuptake inhibitors; sexual function; quality of life; cognition
MeSH Terms: interventions — Hormone Replacement Therapy; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hormone Therapy: Women using hormone replacement therapy (estrogen only or oestrogen and progestin) for treating climacteric symptoms.
  Interventions: Drug: Hormone replacement therapy
- Selective Serotonin Reuptake Inhibitors: Women using selective serotonin reuptake inhibitors for treating climacteric symptoms.
  Interventions: Drug: Selective serotonin reuptake inhibitors
- Control Group: Women not using hormone replacement therapy or selective serotonin reuptake inhibitors

INTERVENTIONS:
Drug: Hormone replacement therapy — Hormone replacement therapy: menopause hormone therapy with estrogen-only or oestrogen-progestin.
  Groups: Hormone Therapy
Drug: Selective serotonin reuptake inhibitors — Selective serotonin reuptake inhibitors: anyone in the category, e.g.: fluoxetine, sertraline, etc.
  Groups: Selective Serotonin Reuptake Inhibitors

SUMMARY:
Cross-sectional study with postmenopausal women using hormone therapy or serotonin reuptake inhibitor to relieve climacteric symptoms or without any treatment. Participants will answer three questionnaires: FSFI (the Female Sexual Function Index), MENQOL (Menopause-specific Quality of Life) and MEEM (Mini-Mental State Examination). The results will be compared according to treatment group.

DETAILED DESCRIPTION:
Climacteric is a period marked by the reduction of estrogen levels, which leads to the occurrence of various symptoms that can affect a woman's physical, mental, sexual health and quality of life. The use of hormonal therapy (HT), with replacement of estrogen or estrogen and progestin, is indicated to alleviate these symptoms, aiming to improve the woman's quality of life. In addition, it is possible to use other forms of treatment to alleviate these symptoms, including selective serotonin reuptake inhibitors (SSRI), which play a major role in vasomotor symptoms. SSRIs have been used with moderate success in women who have contraindications to the use of HT or do not wish to use it. Objective: This study aims to analyze and compare the effects of HT and SSRIs in the treatment of climacteric symptoms in relation to cognitive and sexual function and quality of life in climacteric women. Methodology: This is a cross-sectional study to be carried out with menopausal women treated at the Centro de Atenção Integral à Saúde da Mulher (CAISM) in the city of São Bernardo do Campo/SP/Brazil. Participants who sign the Informed Consent Form will answer 3 questionnaires: FSFI (Female Sexual Function Index), WHOQOL-Bref (World Health Organization Quality of Life Instrument Bref) and MEEM (Mini-Mental State Examination). The results will be compared according to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged between 45 and 65 years who are literate;
* Patients with at least 6 months of follow-up at the institution and who consented to participate in the research.

Exclusion Criteria:

* Women with psychiatric illness;
* Being on medication with action on the Central Nervous System due to psychiatric indication;
* Cognitive impairment that makes it impossible to understand the issues;
* Illiteracy;
* Absence of at least one sexual activity in the last 4 weeks.

Ages: 45 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged between 45 and 65 years who are literate treated with hormone replacement therapy or selective serotonin reuptake inhibitors for relieve of cllimacteric symptoms, or not yet under any of both treatment.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Score at Female Sexual Function Index scale (DSDI) | Day 1
  Association between treatments and FSFI global score
Score at World Health Organization quality of life assessment - bref scale (WHOQOL-Bref) | Day 1
  Association between treatments and WHOQOL-Bref score
Score at Mini-Mental State Examination scale | Day 1
  Association between treatments and Mini-Mental State Examination score

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pompei, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Centro de Atenção Integral à Saúde da Mulher, São Bernardo do Campo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
This is a small study to know regional data